CLINICAL TRIAL: NCT05263843
Title: Différences de Genre Dans l'Activation Des NET et Son Implication Dans la Formation de Fibrose Cardiaques Chez Les Patients Adultes Avec Une Cardiopathie congénitale Complexe FIBRONETx Gender
Brief Title: Gender Difference in NET Activation in Patients With Congenital Heart Disease and Heart Failure
Acronym: FIBRONETx
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Research Agency, France (Other); European Commission (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211359
Record Dates: First submitted 2022-02-09; First posted 2022-03-03 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Congenital Heart Disease; Heart Failure; Gender
Keywords: Congenital heart disease; Heart failure; Gender; Fibrosis; Inflammation
MeSH Terms: conditions — Heart Defects, Congenital; Heart Failure; Coitus; Fibrosis; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At the end of the study, the samples may be used for further analysis not described in the initial protocol but which may be useful for investigation of congenital cardiopathy in light of advances in scientific knowledge, provided the participant is informed and does not oppose this, as stated in the information note/consent form.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with a complex congenital heart disease
  Interventions: Diagnostic Test: Biological markers of myocardial fibrosis
- controls: healthy subjects
  Interventions: Diagnostic Test: Biological markers of myocardial fibrosis

INTERVENTIONS:
Diagnostic Test: Biological markers of myocardial fibrosis — Blood sample for measurements of NET activation and collagen biomarkers

SUMMARY:
Neutrophil hyperactivation has detrimental effects on cardiac tissue after injuries, leading to fibrosis lesions and cardiac dysfunction. It is now well-established that women present with different clinical symptoms in cardiovascular disease compared to men. A cardioprotective effect in women has been suggested in some studies including patients with congenital heart disease (CHD) and heart failure. Our hypothesis is that estrogen protects the hearts of female patients aged 18-45 with CHD. There is no information available as to the involvement of neutrophils in heart failure in females compared to male patients, and therefore this study will provide important information for both the CHD and neutrophil biology fields comparing NET activation in women and men with severe CHD.

DETAILED DESCRIPTION:
100 patients (50 men and 50 women including 25% with a history of pregnancy) aged 18-45 years with moderate and severe CHD (Fallot, systemic RV, and single ventricle), where fibrosis has been identified as a risk factor for heart failure, will be included. A control group of 50 patients (25 men and 25 women) were matched on age and sex.

The main objective of the study is to study the difference in NET activation between men and women with complex congenital heart disease.

Secondary objectives are:

* To compare the NET activity between healthy subjects vs. patients at inclusion.
* To compare male vs. female NET activity in healthy subjects at inclusion.
* To study the existence of associations of NET with biomarkers of fibrosis (biological and imaging) at baseline in men and women with complex congenital heart disease.
* To study the protective value of pregnancy on inflammatory mechanisms and the formation of fibrosis involved in impaired ventricular function and heart failure in these patients.

The enrolled patients will have blood samples collected for analysis of PAD4/NETs biomarkers, and fibrosis markers. NET/fibrosis markers will be correlated with clinical/laboratory parameters, notably NET/PAD4 levels with markers of fibrosis such as collagen biomarkers, ECG, echocardiographic, and cardiac magnetic resonance imaging biomarkers.

ELIGIBILITY:
Inclusion Criteria:

Patients:

Male or female aged 18 to 45; having one of the following 3 complex congenital heart disease:

Congenital heart disease with a systemic right ventricle Congenital heart disease with a single ventricle palliated by Fontan's circulation Tetralogy of Fallot repaired - Patient benefiting from a social security scheme or having rights, or CMU; obtaining informed consent from the patient

Healthy subjects:

Age over 18 years old, matched by sex and age +/- 5 years; Normal ECG; with a prior clinical examination; benefiting from social security; obtaining informed consent from the patient

Exclusion Criteria:

Patients:

patients with cyanosis defined as saturation ≤ 90% at rest; Usual MRI contraindications Possible confounding factors with increased NET formation unrelated to thrombosis, namely cancer, rheumatoid arthritis, lupus, antiphospholipid syndrome, history of pre-Eclampsia or hypertension; Contraindication to performing a stress test; Glomerular filtration rate <30ml / min / 1.73m² of body surface area A physical or mental disability that does not allow for a stress test; Pregnant or lactating patient;Patient under legal protection

- Healthy subjects: Known or detectable history of a heart attack on the ECG; known or detectable primary or secondary cardiomyopathy on ECG; history of chest radiation therapy or chemotherapy;Possible confounding factors with increased NET formation unrelated to thrombosis, namely cancer, rheumatoid arthritis, lupus, antiphospholipid syndrome, history of pre-Eclampsia or hypertension Contraindication to performing a stress test;Glomerular filtration rate <30ml / min;BMI>30; Pregnant or lactating patient;Patient under legal protection

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 50 male and 50 female including half of them with a history of pregnancy
Study Population: The study population will therefore be represented by:
  * heart diseases at risk of heart failure with an equal proportion of men and women to be able to study the protective character of the female sex on the inflammatory process and the development of myocardial fibrosis.
  * healthy adult subjects.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2025-02-23 (Estimated); Study Completion 2025-02-23 (Estimated)

PRIMARY OUTCOMES:
NET activation levels and PAD4 Levels | baseline
  Measurements of MPO-DNA, citrullinated histone, Elastase, Calprotectine, MMP9, NGAL, and MPO, IL-8

SECONDARY OUTCOMES:
The association of NET / PAD4 biomarker levels will be analyzed to NYHA functional class. | baseline
  The association between NYHA functional class (I, II, III and IV) and the following measurements will be analyzed:
  * MPO-DNA (UA/mL)
  * Citrullinated histone (optic density unit)
  * Elastase (pg/mL)
  * Calprotectine (pg/mL)
  * MMP9 (pg/mL)
  * NGAL (pg/mL)
  * MPO (UA/mL)
  * IL-8 (pg/ml)
The association of NET / PAD4 biomarker levels will be analyzed in relation to QRS width and late potentials. | baseline
  The association between each ECG parameters: QRS width (ms) and late potentials (present or absent) and the following measurements will be analyzed:
  * MPO-DNA (UA/mL)
  * Citrullinated histone (optic density unit)
  * Elastase (pg/mL)
  * Calprotectine (pg/mL)
  * MMP9 (pg/mL)
  * NGAL (pg/mL)
  * MPO (UA/mL)
  * IL-8 (pg/ml)
The association of NET / PAD4 biomarker levels will be analyzed in relation to ventricular function, ventricular longitudinal strain, diastolic parameters, presence of valvular disease, change in systemic ventricular filling profile after exercise | baseline
  The association between each echographic measurement: ventricular function, ventricular longitudinal strain, diastolic parameters, presence of valvular disease, change in systemic ventricular filling profile after exercise and the following measurements will be analyzed:
  * MPO-DNA (UA/mL)
  * Citrullinated histone (optic density unit)
  * Elastase (pg/mL)
  * Calprotectine (pg/mL)
  * MMP9 (pg/mL)
  * NGAL (pg/mL)
  * MPO (UA/mL)
  * IL-8 (pg/ml)
The association of NET / PAD4 biomarker levels will be analyzed in relation to measurement of myocardial stiffness. | baseline
  The association between myocardial stiffness (in KPa, measured with ultrafast cardiac echography) and the following measurements will be analyzed :
  * MPO-DNA (UA/mL)
  * Citrullinated histone (optic density unit)
  * Elastase (pg/mL)
  * Calprotectine (pg/mL)
  * MMP9 (pg/mL)
  * NGAL (pg/mL)
  * MPO (UA/mL)
  * IL-8 (pg/ml)
The association of NET / PAD4 biomarker levels will be analyzed in relation to volumes, masses and ventricular ejection fraction, late enhancement and T1 measurement | baseline
  The association between each parameters of cardiac magnetic resonance imaging: volumes, masses and ventricular ejection fraction, late enhancement and T1 measurement and the following measurements will be analyzed :
  * MPO-DNA (UA/mL)
  * Citrullinated histone (optic density unit)
  * Elastase (pg/mL)
  * Calprotectine (pg/mL)
  * MMP9 (pg/mL)
  * NGAL (pg/mL)
  * MPO (UA/mL)
  * IL-8 (pg/ml)
The association of NET / PAD4 biomarker levels will be analyzed in relation to biological markers: BNP, CRPus, troponin, biomarkers of collagen metabolism. | baseline
  The association between each biological markers: BNP (pg/ml), CRPus (mg/L), troponin (ng/L), biomarkers of collagen metabolism (PICP (ng/Ml), P3NP (ng/ml), ICTP (microgr/L), MMP1 (ng/ml), TIMP1 (ng/ml), galactine 3 (ng/ml)) and the following measurements will be analyzed :
  * MPO-DNA (UA/mL)
  * Citrullinated histone (optic density unit)
  * Elastase (pg/mL)
  * Calprotectine (pg/mL)
  * MMP9 (pg/mL)
  * NGAL (pg/mL)
  * MPO (UA/mL)
  * IL-8 (pg/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Magalie Ladouceur, Pr, Principal Investigator — Hôpital Européen Georges-Pompidou
Locations (2):
- France (2):
  - C01 - Hôpital Européen Georges Pompidou - Unité des cardiopathies congénitales de l'adulte, Paris
  - C02- Hôpital Européen Georges Pompidou - CIC, Paris

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered.
  Data sharing must respect the agreements made with funders.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractual agreement.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).

REFERENCES:
- [Background] Marelli AJ, Mackie AS, Ionescu-Ittu R, Rahme E, Pilote L. Congenital heart disease in the general population: changing prevalence and age distribution. Circulation. 2007 Jan 16;115(2):163-72. doi: 10.1161/CIRCULATIONAHA.106.627224. Epub 2007 Jan 8. PMID 17210844
- [Background] Burchill LJ, Broberg CS, Maxwell BG, McLarry J, Opotowskuy S. National Heart Failure Admissions and Associated Mortality Trends in Adults With Congenital Heart Disease in the United States, 1998-2011. J Heart Lung Transplant. 1 avr 2015;34(4):S155.
- [Background] Moussa NB, Karsenty C, Pontnau F, Malekzadeh-Milani S, Boudjemline Y, Legendre A, Bonnet D, Iserin L, Ladouceur M. Characteristics and outcomes of heart failure-related hospitalization in adults with congenital heart disease. Arch Cardiovasc Dis. 2017 May;110(5):283-291. doi: 10.1016/j.acvd.2017.01.008. Epub 2017 Mar 14. PMID 28314706
- [Background] Diller G-P. Incidence and Prevalence of Heart Failure in Adults with Congenital Heart Disease. In: Swan L, Frogoudaki AA, éditeurs. Heart Failure in Adult Congenital Heart Disease [Internet]. Cham: Springer International Publishing; 2018. p. 3-9. (Congenital Heart Disease in Adolescents and Adults). Disponible sur: https://doi.org/10.1007/978-3-319-77803-7_1
- [Background] Khairy P, Fernandes SM, Mayer JE Jr, Triedman JK, Walsh EP, Lock JE, Landzberg MJ. Long-term survival, modes of death, and predictors of mortality in patients with Fontan surgery. Circulation. 2008 Jan 1;117(1):85-92. doi: 10.1161/CIRCULATIONAHA.107.738559. Epub 2007 Dec 10. PMID 18071068
- [Background] Engelings CC, Helm PC, Abdul-Khaliq H, Asfour B, Bauer UM, Baumgartner H, Kececioglu D, Korten MA, Diller GP, Tutarel O. Cause of death in adults with congenital heart disease - An analysis of the German National Register for Congenital Heart Defects. Int J Cardiol. 2016 May 15;211:31-6. doi: 10.1016/j.ijcard.2016.02.133. Epub 2016 Mar 2. PMID 26970963
- [Background] Diller GP, Kempny A, Alonso-Gonzalez R, Swan L, Uebing A, Li W, Babu-Narayan S, Wort SJ, Dimopoulos K, Gatzoulis MA. Survival Prospects and Circumstances of Death in Contemporary Adult Congenital Heart Disease Patients Under Follow-Up at a Large Tertiary Centre. Circulation. 2015 Dec 1;132(22):2118-25. doi: 10.1161/CIRCULATIONAHA.115.017202. Epub 2015 Sep 14. PMID 26369353
- [Background] Zomer AC, Vaartjes I, van der Velde ET, de Jong HM, Konings TC, Wagenaar LJ, Heesen WF, Eerens F, Baur LH, Grobbee DE, Mulder BJ. Heart failure admissions in adults with congenital heart disease; risk factors and prognosis. Int J Cardiol. 2013 Oct 3;168(3):2487-93. doi: 10.1016/j.ijcard.2013.03.003. Epub 2013 Apr 18. PMID 23602867
- [Background] Wang F, Liu A, Brophy JM, Cohen S, Abrahamowicz M, Paradis G, Marelli A. Determinants of Survival in Older Adults With Congenital Heart Disease Newly Hospitalized for Heart Failure. Circ Heart Fail. 2020 Aug;13(8):e006490. doi: 10.1161/CIRCHEARTFAILURE.119.006490. Epub 2020 Jul 16. PMID 32673500
- [Background] Ghali JK, Krause-Steinrauf HJ, Adams KF, Khan SS, Rosenberg YD, Yancy CW, Young JB, Goldman S, Peberdy MA, Lindenfeld J. Gender differences in advanced heart failure: insights from the BEST study. J Am Coll Cardiol. 2003 Dec 17;42(12):2128-34. doi: 10.1016/j.jacc.2003.05.012. PMID 14680739
- [Background] Zomer AC, Ionescu-Ittu R, Vaartjes I, Pilote L, Mackie AS, Therrien J, Langemeijer MM, Grobbee DE, Mulder BJ, Marelli AJ. Sex differences in hospital mortality in adults with congenital heart disease: the impact of reproductive health. J Am Coll Cardiol. 2013 Jul 2;62(1):58-67. doi: 10.1016/j.jacc.2013.03.056. Epub 2013 May 1. PMID 23644083